CLINICAL TRIAL: NCT04055584
Title: PCR Techniques of Dried Sputum Using a Spotcard
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Onno Akkerman, Principal Investigator, University Medical Center Groningen
Other Study IDs: PCR techniques of dried sputum
Record Dates: First submitted 2019-08-06; First posted 2019-08-14 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — Sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sputum spot
  Interventions: Diagnostic Test: Sputum

INTERVENTIONS:
Diagnostic Test: Sputum — DNA extraction and perform a diversity of molecular diagnostic tests

SUMMARY:
Molecular testing for mutations in M. tuberculosis genes associated to resistance of anti tuberculosis (TB) drugs is already part of standard laboratory TB diagnostic.

This implicates earlier knowledge of possible resistance and thus prevents unnecessary treatment and the chance of treatment failure or treatment related toxicity.

The molecular laboratory diagnostics is widely spread in high income, low TB endemic countries. However, the low income countries lack widespread facilities to test for susceptibility, either genotypic or phenotypic. Performing molecular diagnostics on sputum collected with a spot card could improve accessibility to molecular testing.

This study examines if sputum collected and put on spot cards could be used for multiple molecular tests for the detection, identification and susceptibility prediction of TB. This means that DNA extraction of the sputum from the spot card should be feasible.

The study is a pilot study with adult patients of the tuberculosis department of University Medical Centre Groningen (UMCG) Beatrixoord, Haren as subjects. The sputum produced will be collected, dried on spot cards, and DNA extraction from the card will be tested. If molecular detection is positive for the tuberculosis bacteria additional tests will be performed. Based on the present/absent of mutations in the genes associated to resistance susceptibility can be preditec, different molecular techniques will be performed to identify possible mutations. Furthermore, sputum will be collected as patients produce so. Sputum samples with low bacterial load can be tested as well and can test the sensitivity of the procedure.

Lastly, techniques like RNA detection will be tested to identify the bacterial load. This can be done if more than one sample of patients were collected.

Subjects will be selected on age, participation in standard TDM and drug use. Demographic parameters will be analysed. Sputum samples will be taken twice a week (on Tuesday and Friday).

ELIGIBILITY:
Inclusion Criteria:

* Patients is 18 years or older
* Pulmonary TB confirmed by culture or molecular test
* Producing sputum
* Signed informed consent

Exclusion Criteria:

* Extrapulmonary TB
* Pulmonary TB without production of sputum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary tuberculosis producing sputum
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2019-07-02 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Is it possible to perform a diversity of molecular diagnostic TB tests and in addition new next generation sequencing approaches, with the DNA from the dried sputum spots? | 6 months
  Is it possible to perform a diversity of molecular diagnostic TB tests and in addition new next generation sequencing approaches, with the DNA from the dried sputum spots?

SECONDARY OUTCOMES:
Can we use DNA detection of the sputum from the dried card to certify that in the final utilisation format both the sputum and blood (not collected or tested in this study) are from the same patient? | 6 months
  Can we use DNA detection of the sputum from the dried card to certify that in the final utilisation format both the sputum and blood (not collected or tested in this study) are from the same patient?

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No